CLINICAL TRIAL: NCT03772847
Title: Ginkgolide With Intravenous Alteplase Thrombolysis in Acute Ischemic Stroke Neurological Improving Trial
Acronym: GIANT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Dongyang People's Hospital (Other); Haiyan People's Hospital (Unknown); The Second Affiliated Hospital of Jiaxing University (Other); Tongxiang Second People's Hospital (Unknown); Tongxiang First People's Hospital (Unknown); Changxing People's Hospital (Other); The Central Hospital of Lishui City (Other); The First People's Hospital of Huzhou (Other); Taizhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yan 2018-015
Record Dates: First submitted 2018-09-05; First posted 2018-12-11 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-07

CONDITIONS: Intravenous Alteplase Thrombolysis; Neurological Improving
MeSH Terms: interventions — Ginkgolides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ginkgolide group (Experimental): ginkgolide plus alteplase
  Interventions: Drug: ginkgolide
- control (No Intervention): alteplase

INTERVENTIONS:
Drug: ginkgolide — ginkgolide plus alteplase
  Arms: ginkgolide group

SUMMARY:
Previous clinical studies have confirmed that revascularization or recanalization rate after intravenous thrombolysis is closely related to the formation of thrombus, which also results in poor neurological function after thrombolysis. Platelet activating factor (PAF) strong platelet aggregation may be involved in thrombosis. Formation process. The main components of Ginkgolide injection (Ginkgo) are ginkgolide, ginkgolides A, ginkgolides B and ginkgolides C. Ginkgo biloba lactone can antagonize PAF and has strong anti-platelet aggregation. . Therefore, it can be speculated that ginkgolides injection combined with alteplase intravenous thrombolysis may improve the recanalization rate after thrombolysis and reduce the reocclusion rate.

In addition, clinical studies have also found that ginkgolide injection has a good auxiliary effect on hypertensive intracerebral hemorrhage, which can regulate inflammatory factors such as IL-6, TNF-α and high-sensitivity C-reactive protein (CRP) in patients. Recovery of neurological function in patients. It is well known that TNF-α, IL-β, IL-1, IL-6, IFN-γ, etc. are all inflammatory factors associated with reperfusion injury. Therefore, we speculate that ginkgolides injection may also regulate inflammatory factors associated with reperfusion injury, such as IL-6, TNF-α, thereby reducing reperfusion injury, thereby improving patient prognosis.

The aim of this study was to determine the clinical efficacy of ginkgolides injection combined with alteplase in the treatment of acute ischemic stroke, and to improve the prognosis of patients with thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old, clinically diagnosed as acute ischemic stroke;
2. in accordance with the indications for intravenous thrombolysis;
3. The patient or family member signs an informed consent form.

Exclusion Criteria:

1. Patients with transient ischemic attack;
2. Imaging examination of patients with cerebral hemorrhage
3. patients with cerebral arteritis
4. ALT, AST ≥ 3 times the upper limit of normal value, Cr ≥ 1.5 times the upper limit of normal value
5. There is a tendency to bleed, and severe bleeding has occurred within 3 months
6. Patients with ginkgo drugs, alcohol, glycerol allergies or allergies
7. Patients with pregnancy plans, pregnancy and breastfeeding
8. Patients who participated in other drug clinical studies in the past month
9. Patients considered by the investigator to be unfit to participate in the clinical study (eg, mental, abnormal, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a 90-day modified Rankin Scale (mRS) score below 2 | 90 days
  mRS 0-6, higher indicate worse outcome

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale(NIHSS) scores between the two groups at baseline, 24 hours, 7 days, and 14 days | 14 days
  NIHSS 0-42, and higher indicate worse outcome
recurrence rate of cerebrovascular disease in 1-month and 3-month follow-up | 3 months
incidence of compound events (include cerebrovascular events,myocardial infarction, angina pectoris, and systemic embolism） | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ze Xin Chen, Study Chair — 2nd affiliated hospital of Zhejiang University，School of Medicine
Locations (1):
- Min Lou, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang X, Zhong W, Ma X, Zhang X, Chen H, Wang Z, Lou M. Ginkgolide With Intravenous Alteplase Thrombolysis in Acute Ischemic Stroke Improving Neurological Function: A Multicenter, Cluster-Randomized Trial (GIANT). Front Pharmacol. 2021 Dec 3;12:792136. doi: 10.3389/fphar.2021.792136. eCollection 2021. PMID 34925044